CLINICAL TRIAL: NCT01667939
Title: A Supervised Nutritional Program in Pregnancies Diminish the NF-κB Expression in Placenta
Brief Title: A Supervised Nutritional Program in Pregnancies and NF-κB Expression in Placenta
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Materno-Perinatal Hospital of the State of Mexico (Other)
Collaborators: National Council of Science and Technology, Mexico (Other); Secretariat of Public Education (SEP) (Unknown)
Responsible Party: Principal Investigator, Hugo Mendieta Zeron, General Internal Medicine, Researcher, Materno-Perinatal Hospital of the State of Mexico
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HMPMP05/06/09
Record Dates: First submitted 2012-08-15; First posted 2012-08-17 (Estimated); Last update posted 2012-08-17 (Estimated); Status verified 2012-08

CONDITIONS: Dietary Habits
Keywords: adequacy; diet; pregnancy
MeSH Terms: conditions — Feeding Behavior | interventions — Diet, Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- pregnancy diet (Experimental): Healthy Eating Index (HEI) in supervised pregnancies
  Interventions: Behavioral: Healthy Eating Index (HEI) in supervised pregnancies
- unsupervised pregnancy (No Intervention): women attending the obstetrics unit who did not follow a supervised diet

INTERVENTIONS:
Behavioral: Healthy Eating Index (HEI) in supervised pregnancies — Dietetic treatment was calculated according to height, weeks of gestation and weight, considering an energy intake of 30 kcal/kg of expected weight, distributing the resulting energy according to the percentage of macronutrients' adequation (55-65% carbohydrates, 10-20% fat and the remainder as proteins).16 On each nutritional visit, 24 hour dietary recall was done and analyzed using NutriKcal®VO software in order to evaluate the Healthy Eating Index (HEI), which is commonly employed to assess pregnant women's dietary adequacy (on a scale from 0-100), through the consumption of 12 components of food groups described previously. An improvement in diet was considered when the initial HEI score improved more than one point during the next nutritional assessment.
  Other Names: NutriKcal®VO software
  Arms: pregnancy diet

SUMMARY:
Nuclear factor kappa B (NF-κB) pathway and oxidative stress participate in endothelial dysfunction, which is one of the causes of preeclampsia. Among the human antioxidant mechanisms there are the enzymes catalase (CAT), glutathione peroxidase (GPx) and superoxide dismutase (SOD). Our aim was to measure NF-κB and oxidative stress in pregnant women submitted to an individualized diet during pregnancy.

DETAILED DESCRIPTION:
Obesity during pregnancy is associated with exaggerated metabolic adaptation, endothelial dysfunction and an increased risk of adverse pregnancy outcomes, including preeclampsia, a major cause of maternal and fetal morbidity and mortality characterized by increased blood pressure, proteinuria and edema, which affects approximately 3% to 7% of all pregnant women. Other risk factors, besides obesity, that increase the likelihood of developing preeclampsia include chronic hypertension, and diabetes mellitus.

Reactive oxygen species (ROS) [superoxide anions (•O2-), hydrogen peroxide (H2O2) and hydroxyl radicals (•OH)],5 interact with proteins, nucleic acids and lipids and in a process called lipid peroxidation (LPO), can cause severe cell and tissue damage. There is current evidence that ROS are common activators of nuclear factor-kappa B (NF-κB), a factor that initiates a systemic inflammatory process by promoting the synthesis of cytokines, interleukin (IL)-6, IL-8, monocyte chemotactic protein-1 (MCP-1) and expression of intercellular adhesion molecule (ICAM-1).

To maintain balance of the oxidative state, the human body possesses intracellular antioxidant enzyme systems, including superoxide dismutase (SOD, glutathione peroxidase (GPx), and catalase (CAT), which is located mainly in peroxisomes and cytoplasm of the cell.

The epidemiology of preeclampsia, which is more common among poor women, had previously suggested that nutrients may be involved in the disorder, unfortunately, the nutritional data obtained from women with the syndrome has been poorly defined.

The objective of this paper was to provide an overview of the biological plausibility and potential mechanisms underlying associations among maternal nutrition, oxidative stress in placenta and the risk of preeclampsia.

ELIGIBILITY:
Inclusion Criteria:

* Women in their first trimester of pregnancy

Exclusion Criteria:

* multiple pregnancies
* prior history of chronic-metabolic diseases

Ages: 18 Years to 36 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2009-06; Primary Completion 2010-12 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Placental expression of NF-κB | two years
  measure of gene expression by real time PCR

CONTACTS AND LOCATIONS:
Overall Officials: Hugo Mendieta Zeron, PhD, Principal Investigator — Materno-Perinatal Hospital "Monica Pretelini"
Locations (1):
- Materno-Perinatal Hospital "Mónica Pretelini", Toluca, State of Mexico, Mexico